CLINICAL TRIAL: NCT00347048
Title: Tacrolimus (FK506) P-III Placebo-Controlled Double-Blind Study in Moderate to Severe Refractory Ulcerative Colitis Patients
Brief Title: Tacrolimus (FK506) Study in Moderate to Severe Refractory Ulcerative Colitis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F506-CL-1107
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; tacrolimus; FK506; treatment outcome
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tacrolimus
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tacrolimus — oral
  Other Names: FK506; Prograf
  Arms: 1
Drug: Placebo — oral
  Arms: 2

SUMMARY:
This study consists of a 2-week placebo-controlled double-blind inter-group efficacy study in moderate to severe refractory ulcerative colitis (UC) patients followed by a maximum of 12-week open-label efficacy and safety study in responders.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe refractory UC patients
* Disease activity: more than 4 times of stool a day, bloody stool, moderate to severe endoscopic finding
* Steroid resistance or dependence to meet at least one of the following condition:no efficacy with more than 40mg/day or 1mg/kg/day of steroid over at least 1 week, no efficacy with 30-40mg/day of steroid over at least 2 weeks,exacerbation along with steroid reduction

Exclusion Criteria:

* Mild or fulminant type
* Renal failure patients, hepatic failure patients
* Patients taking 6-mercaptopurine, cyclosporin or other immunosuppressants within 12 weeks prior to entry
* Patients who received LCAP or GCAP within 2 weeks prior to entry
* Patients who changed the dose of steroid or started steroid within 2 weeks prior to entry.
* Patients who changed the dose of steroid or started steroid within 1 week prior to entry in case they received more than 40 mg/ day or 1mg/kg/day of steroid just before the study.

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Improvement of Disease activity index score (DAI score) | 2 Weeks

SECONDARY OUTCOMES:
Changes of DAI score ( Total & each item) | 2 Weeks
Changes of clinical severity and symptom | 2 Weeks
Endoscopic finding | 2 Weeks
Patients impression | 2 Weeks
Amount of steroid | 2 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (6):
- Japan (6):
  - Chubu Region
  - Hokkaido Region
  - Kansai Region
  - Kanto Region
  - Kyushu Region
  - Shin'etsu Region